CLINICAL TRIAL: NCT07014553
Title: Effect of Web-based Nursing Navigator Programme on Breast Cancer Screening Behaviors in Women at High Risk of Breast Cancer
Acronym: WeT-HNP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Tuğçe çiçekli taşdemir, Lecturer, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IUC-NURSE-TÇT-01
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer Risk
Keywords: breast cancer; nursing; public health nursing; web based; nursing navigator programme
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 6-week web-based nursing navigation programme
  Interventions: Behavioral: web based nursing navigator programme
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: web based nursing navigator programme — health education guidance surveillance case management
  Arms: Experimental group

SUMMARY:
The aim of this project is to determine the effect of the Web-Based Nurse Navigation Program on breast cancer screening behaviors (mammography, BSE, CBE) in women at high risk of breast cancer. The program to be developed within the scope of the project is named as "Web-Based Nurse Navigation Program (WeT-HNP)", which reflects the web-based and navigation concepts.

DETAILED DESCRIPTION:
Breast cancer is a very important health problem affecting women's health in the world and in our country. It was reported that 685,000 people died of breast cancer in the world in 2020. The American Cancer Society estimates that approximately 310,720 new cases of invasive breast cancer will be detected in women in the United States in 2024, approximately 56,500 new cases of ductal carcinoma in situ (DCIS) will be detected, and approximately 42,250 women will die from breast cancer. In Turkey, breast cancer is the most common type of cancer in women and the cause of most deaths. In national reports for our country, it was reported that the frequency of breast cancer in women in 2018 was 48.6 per hundred thousand and the number of newly diagnosed patients in the same year was 22,500. Early diagnosis of breast cancer, which is a very important health problem in terms of women's health, reduces mortality and provides the opportunity for breast-conserving surgery. Today, the most effective approach in reducing mortality rates in breast cancer is early diagnosis/screening methods. Early diagnosis/screening methods aim to detect abnormal changes in women's breast tissue at an early stage. Breast self-examination (BSE), clinical breast examination (CBE) and mammography are widely recommended early diagnosis/screening methods for the early detection of breast cancer. In order to detect breast cancer at the earliest stage, it is recommended that women without symptoms in our country have a BSE every month starting at the age of 20, have a CBE once a year, and have a mammogram every 2 years between the ages of 40-69.It is recommended that women at high risk of breast cancer start breast cancer screening earlier and be monitored more frequently than women without symptoms. The American Cancer Society recommends that women at high risk of breast cancer have a mammogram every year after the age of 30.

ELIGIBILITY:
Inclusion Criteria:

* Being 30-70 years old,
* Not having been diagnosed with breast cancer,
* Not having been included in a breast health program before,
* Not having had a mammogram in the last year,
* Being at high risk of breast cancer according to the Tyrer-Cuzick Model,
* Having a phone, computer or laptop with internet access,
* Not having a health problem that prevents vision or hearing,
* Being willing to participate in the study.

Exclusion Criteria:

* Not being able to read or write,
* Having a history of breast cancer,
* Not being at high risk of breast cancer,
* Being pregnant or postpartum,
* Not agreeing to participate in the study.

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
mammography rates | baseline, 6 months
  browsing behavior monitoring form
rate of breast self-examination | baseline, 3 months
  screening behaviors follow-up form
rate of clinical breast examination | baseline, 6 months
  screening behaviors follow-up form

SECONDARY OUTCOMES:
Health perceptions | baseline, 6 months
  Breast Cancer Health Belief Model Scale Results
Breast cancer fear score | baseline, 6 months
  Breast Cancer Fear Scale
perception of mammography competence | baseline, 6 months
  Mammography Competence Scale

CONTACTS AND LOCATIONS:
Overall Officials: Selda Seçginli, Prof. Dr., Study Director — Atlas University
Locations (2):
- Turkey (Türkiye) (2):
  - Cancer early diagnosis screening and education center, Istanbul, Büyükçekmece
  - Family health center, Istanbul, Büyükçekmece

IPD SHARING:
Plan to Share IPD: No